CLINICAL TRIAL: NCT03660982
Title: Familial Aggregation and Biomarkers in REM Sleep Behaviour Disorder: a Case-control Family Study
Brief Title: Familial Aggregation and Biomarkers in REM Sleep Behaviour Disorder.
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Dr. Zhang Jihui, Assistant professor, Chinese University of Hong Kong
Other Study IDs: 12131501
Record Dates: First submitted 2018-08-30; First posted 2018-09-07 (Actual); Last update posted 2021-08-06 (Actual); Status verified 2021-08

CONDITIONS: REM Sleep Behavior Disorder
MeSH Terms: conditions — REM Sleep Behavior Disorder

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — TFT-SEP Serum Clot, Vitamin B12-SEP Serum clot, Folate- SEP Serum clot, CBC-EDTA, Fasting Glucose-Fluoride

GROUPS / COHORTS (2):
- FDRs of RBD cases: FDRs of RBD cases. The diagnosis of RBD is based on ICSD-II criteria, as confirmed by v-PSG and with the aid of REM sleep behaviour disorder questionnaire (RBDQ-HK). RBD cases which are secondary to narcolepsy, neurodegenerative diseases or other neurological diseases are excluded.
- FDRs of non-RBD controls: FDRs of non-RBD controls. Non-RBD control probands are free of narcolepsy, significant clinical RBD symptoms and other neurological diseases.

SUMMARY:
In this cohort study, the investigators aim to study the familial aggregation of REM sleep behavior disorder (RBD) and compare the differences in major biomarkers of neurodegeneration, including percentage of EMG activity during REM sleep, cognitive functions, autonomic dysfunction, and psychiatric disorders, between unaffected first degree relatives of RBD cases and non-RBD controls.

DETAILED DESCRIPTION:
REM sleep behavior disorder (RBD) is a parasomnia characterized by abnormal behavioral manifestations during REM sleep. Previous case-control studies and prospective studies have documented the progression of α-synucleinopathy neurodegeneration in relation to RBD and have identified some biomarkers of predicting neurodegeneration in patients with iRBD, such as olfactory dysfunction, color vision deficit, autonomic dysfunction, tonic EMG activity during REM sleep, and psychiatric disorder. However, these biomarkers might precede the onset of RBD, as a result, searching for biomarkers for the neurodegeneration before RBD onset is helpful to map the progression of neurodegeneration. In this regard, the investigators aim to study the familial aggregation of RBD and its core features, and compare the differences in major biomarkers of neurodegeneration, including percentage of EMG activity during REM sleep, cognitive functions, autonomic dysfunction, and psychiatric disorders, between unaffected first degree relatives of RBD cases and non-RBD controls.

ELIGIBILITY:
Inclusion Criteria:

1. Chinese aged 40 or above;
2. Being capable of giving informed consent for participation of the study;
3. Sex matched between relatives from probands and controls.

Exclusion Criteria:

1. Aged 39 or below;
2. Not capable of giving informed consent for participation of the study

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: We established a case-control cohort of RBD with regular follow-ups and we have now accumulated over 280 RBD cases and age-sex matched controls. Proband of RBD and non-RBD controls will be recruited from this cohort. The control probands were initially recruited from the community and clinical samples (those with other sleep disorders such as obstructive sleep apnea syndrome) that did not have RBD as confirmed by clinical and vPSG assessments.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2014-10-01; Primary Completion 2022-09-30 (Estimated); Study Completion 2022-09-30 (Estimated)

PRIMARY OUTCOMES:
The prevalence rate of probable RBD among first degree relatives of RBD probands | 15 minutes
  The prevalence rate of probable RBD based on the self-reported/proxy-reported RBD symptoms in RBDQ-HK among first degree relatives of RBD probands in comparison to that of first degree relatives of controls.
The weighted prevalence rate of confirmed RBD among first degree relatives of RBD probands. | one night (8 hours)
  The weighted prevalence rate of first degree relatives meeting full ICSD-II2 diagnostic criteria for RBD confirmed by clinical history and vPSG.

SECONDARY OUTCOMES:
The percentage of REM-related EMG activity (REMREEA) | one night (8 hours)
  The percentage of REM-related EMG activity (REMREEA) is the most reliable and valid marker in differentiating patients with RBD from normal controls. Basically, the REMREEA include two components, namely phasic EMG activity and tonic EMG activity, respectively. The phasic EMG events were defined as any burst of EMG activity lasting 0.1 to 5 sec with amplitude > 4 times the background EMG activity and will be score on the basis of 3-second mini-epoch during REM sleep. Each 30-sec epoch during REM sleep was scored as tonic or atonic depending on whether tonic chin EMG activity was present for more or less than 50% of the epoch. The total EMG activity was presented as the percentage of REM related EMG activity (REMREEA) with the percentage of tonic EMG activity plus the percentage of phasic EMG activity.
Significant motor activity | one night (8 hours)
  Significant motor activity were recorded by video-polysomnography. The motor analysis will be scored according to the previously established method. In view of the potential problem in inter-rater reliability in those mild motor activities, we will only include those complex activities and vocalizations in the analyses. It has been shown that there are large differences in the significant motor activities between patients with RBD and normal controls. In view of the relatively high night-to-night variability and low inter-rater reliability in scoring motor activity, it will be considered as secondary outcome.
Other biomarkers of RBD in the first degree relatives of RBD patients. | 2 hours
  Previous studies have also confirmed that RBD patients present with autonomic dysfunction, olfactory dysfunction, color vision deficit, neurocognitive function, and a higher rate of psychiatric disorders, these markers will also be considered as secondary biomarkers and will be compared in the first degree relatives of between patients and controls.

CONTACTS AND LOCATIONS:
Overall Officials: Jihui Zhang, PhD, Principal Investigator — Chinese University of Hong Kong; Yun Kwok Wing, MBChB, Study Director — Chinese University of Hong Kong; Siuping LAM, Study Director — Chinese University of Hong Kong; Vicent Chung-tong MOK, Study Director — Chinese University of Hong Kong
Locations (1):
- Department of psychiatry, Faculty of Medicine, The Chinese University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Undecided
In this stage, we didn't decide which information of IPD will share with other researchers.